CLINICAL TRIAL: NCT06598787
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 for Injection in Patients With Recurrent Glioblastoma
Brief Title: A Study of BL-B01D1 in Patients With Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-205
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 for Injection (Experimental): Participants receive BL-B01D1 in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1 for Injection

INTERVENTIONS:
Drug: BL-B01D1 for Injection — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507

SUMMARY:
This is an open-label, multicenter, phase II study to evaluate the safety, efficacy, and pharmacokinetic characteristics of BL-B01D1 for Injection in patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old;
4. Recurrent glioblastoma confirmed by pathology after failure of standard treatment;
5. KPS≥60;
6. The expected survival time as judged by the investigator was ≥3 months;
7. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
8. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
9. No blood transfusion, albumin, colony-stimulating factor, any cell growth factor and/or platelet-raising drugs are allowed within 14 days before the first dose of study drug, and the organ function level must meet the requirements;
10. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN;
11. Urine protein ≤2+ or < 1000mg/24h;
12. A pregnancy test must be performed within 7 days before starting treatment for premenopausal women who are likely to have children, the serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, etc., had been used within 4 weeks or 5 half-lives before the first dose, small molecule targeted therapy had been used within 5 days, palliative radiotherapy, modern Chinese medicine preparations approved by NMPA for anti-tumor treatment had been used within 2 weeks;
2. A history of central nervous system hemorrhage/infarction requiring treatment unrelated to antineoplastic drugs within 6 months before enrollment;
3. History of severe heart disease and cerebrovascular disease;
4. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, severe arrhythmia;
5. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
6. Active autoimmune and inflammatory diseases;
7. Other malignant tumors that progressed or required treatment within 5 years before the first dose;
8. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
9. Patients with poor glycemic control or with diabetic gangrene;
10. Patients with a previous history of ILD, or current ILD or ≥G2 radiation pneumonitis, or suspected to have such disease by imaging during screening;
11. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
12. Patients with a history of allergy to recombinant humanized or human-mouse chimeric antibodies or to any of the excipients of BL-B01D1;
13. Received previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
14. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
15. Had a serious infection within 4 weeks before the first dose of study drug; Indications of active pulmonary infection within 2 weeks before the first dose of study drug;
16. Imaging examination indicated that the tumor had invaded or enveloped the large vessels of the chest, neck, and pharynx, except for those that the investigator thought would not affect the patient's enrollment in the drug;
17. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, PHD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China